CLINICAL TRIAL: NCT04235244
Title: The Effect of Three Different Local Cold Applications on Pain and Ecchymosis in Subcutaneous Heparin Injections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Seda CEVHEROĞLU, PhD of Nursing / Senior Instructor Department of Nursing Faculty of Health Sciences, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: IU-C NURSİNG
Record Dates: First submitted 2020-01-16; First posted 2020-01-21 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Pain; Ecchymosis
Keywords: subcutaneous ınjectıon; cold application; pain; ecchymosis; heparin injection
MeSH Terms: conditions — Pain; Ecchymosis

STUDY DESIGN:
Intervention Model Description: It will be determined by simple randomization method which SC injection will be applied to these four regions. According to the results of randomization;
  * Buzzy, a thermomechanical-analgesia device, was placed 30 seconds before the injection in the right upper abdominal region, and the SC injection was applied by sliding the device to the side of the selected region during the injection
  * SC-LMWH injection was applied to the right lower abdominal region without any cold application
  * Local coolant spray was applied to the left upper abdominal region from a distance of 15 cm for 5 seconds and
  * Before and after the application to the left lower abdominal region, the cold application was performed with a cool-pack for 5 minutes.
  The application of 2x0.6cc standard ready-to-use injectable Enoxiparin, which was requested by the physician according to the SC injection application steps, was applied together with the cold application method determined by randomization.
Masking Description: All SC injections, ecchymosis measurements, VAS evaluation and post-injection follow-up will be performed by the researcher. Immediately after injection, pain intensity at 24, 48 and 72 hours and ecchymosis at 24, 48 and 72 hours will be evaluated
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- left lower abdominal region (Experimental): 5 minutes before and after application to the right upper abdominal region. local cold application
  Interventions: Other: ıce battery
- right upper abdominal region (Experimental): Thermomechanical-analgesia device will be operated 30 seconds before the injection in the right lower abdominal region and the device will be injected by sliding the device to the side of the selected region during the injection,
  Interventions: Other: Thermo mechanical device
- left upper abdominal region (Experimental): Coolant spray will be applied to the upper left abdominal region for 15 sec.
  Interventions: Other: local coolant spray
- right lower abdominal region (No Intervention): SC injection will be applied to the left lower abdominal region without any cold application.

INTERVENTIONS:
Other: Thermo mechanical device — The thermomechanical-analgesia device will be placed and operated 30 seconds before the injection into the abdominal area,and injection will be applied by sliding the device to the side of the selected region during the injection,
  Arms: right upper abdominal region
Other: local coolant spray — Coolant spray will be applied to the abdominal area for 5 seconds at a distance of 15 cm.
  Arms: left upper abdominal region
Other: ıce battery — abdominal bölgeye uygulamadan önce ve sonra 5 dk. lokal soğuk uygulama
  Arms: left lower abdominal region

SUMMARY:
The aim of this study was to investigate the effects of three different cold application methods on ecchymosis and pain in the injection site in patients who received DMAH injection from the SC route.

In the Turkish Republic of Northern Cyprus, the research universe will be composed of the patients who underwent DMAH from the SC path in Internal Medicine Service at a State Hospital under the Ministry of Health. The sample will consist of patients who meet the research criteria, who are informed about the purpose of the research, and who are willing to participate after obtaining the permission of the Ethics Committee and institution. The sample will consist of patients who meet the research criteria, who are informed about the purpose of the research, and who are willing to participate after obtaining the permission of the Ethics Committee and institution. The sample size (d=0.785) was found by reference from the article "effect of ice application on ecchymosis formation in patients undergoing subcutaneous anticoagulant therapy" by Küçükgüçlü and Okumu (2010) and the sample size required for 1-β=0.95 (power) in α=0.05 was n = 38.

Patient Data Sheet, SC Road injection tracking chart, Visual Analog scale, Opsite - Flexigrid measurement tool, Mekano-analgesia (Buzzy) device, local coolant spray and acetate Pen will be used for data collection.

Statistical Package for Social Sciences (SPSS) 25.0 software will be used for statistical analysis of research data. If the data set matches the normal distribution, parametric hypothesis tests will be used, and if the data set does not match the normal distribution, nonparametric hypothesis tests will be used.

DETAILED DESCRIPTION:
Thromboembolism is a frequently seen complication in patients who undergo long-term movement restriction and undergo surgical intervention, causing serious consequences such as pulmonary embolism . For this reason, heparin is frequently used for protective or therapeutic purposes in clinical situations where there is a risk of venous thromboembolism or thromboembolytic events . In the 1980s, low molecular weight heparin (LMWH) preparations, often administered subcutaneously (SC), were developed in order to increase the desired effect and reduce the side effects of heparin applications . It is stated in the literature that SC injection applications can be safely injected into the outer-lateral side of the upper arm, anterior aspect of the thigh, under the scapula and abdominal region . However, in the literature, it is emphasized that ecchymosis and hematoma formation is more common in SC LMWH applications, especially in the arm and thigh areas after SC injection. Therefore, in LMWH applications, it is stated that abdominal region is the most reliable injection site because it has thicker SC tissue compared to other parts of the body . In summary studies, it is recommended as the preferred site for LMWH applications due to the excess of SC fat tissue in the abdominal region, its width to allow rotation of the injection site and the lack of muscle activity .

Systemic and local complications may occur due to heparin injection by SC route. The most important local complications are; ecchymosis at the injection site, hematoma formation and local pain formation at the injection site . In this study, the frequency of ecchymosis; Kuz and Uçar (2001) 11.4%, Dursun and Balcı Akpınar (2014) 28.7%, Küçükgüçlü and Okumuş (2010) 31%, Varghese et al. (2006) 36%, Palese (2013) 38%, Yildirim and Atalay (2005) 57%, Zaybak and Khorshid (2008) reported as 64%. These treatment-related complications complicate the use of the damaged area in subsequent injections, adversely affect drug absorption, and cause physical trauma (ecchymosis, hematoma and pain) and changes in body image.

Pain is a subjective experience that can occur in very different qualities and severity. Pain experienced due to injection is generally defined as a condition that occurs as a result of mechanical trauma in the tissue and stimulates the nerve fiber ends with the entry of the needle into the tissue. Due to the presence of pain receptors in SC tissue, patients often experience discomfort and pain during and after LMWH applications. Pain during injection significantly affects the patient's non-compliance to treatment and pain after injection significantly affects the comfort and life activities of the patient by restricting the use of the extremity . One of the methods used to prevent these negative complications is cold applications.

Local cold administration reduces blood flow through vasoconstriction of the arterioles, controls bleeding and reduces ecchymosis and hematoma development . In addition, local cold application provides vasoconstriction in the tissue to which it is applied, slows blood flow and increases the viscosity of the blood, limits edema and inflammatory process, controls bleeding by reducing capillary permability, and reduces pain perception . With this localized sensory effect, attention is directed towards cold from pain, and thus pain is alleviated by the anesthetic effect of cold . In the studies carried out on the subject; It has been reported that 5 minutes of local humid cold application after SC injection results in a reduction in the severity and pain rate of ecchymosis . Küçükgüçlü and Okumuş (2010); SC indicated that two minutes of ice application to the heparin administration site before and after administration was an effective method of reducing ecchymosis and hematoma. Avşar and Kaşıkçı (2013); They found that two minutes of cold application to the SC injection site reduced ecchymosis and pain. Şendir et al. (2015) SC injection time of 30 seconds and 5 minutes before and after the injection of local ice application, effective in reducing the intensity of pain and ecchymosis was reported to be effective. Similarly, Korkmazcan (2016) emphasizes that application of local ice to the skin is effective for reducing ecchymosis, hematoma and pain in SC LMWH injections. In addition, it is reported that pre-injection coolant spray and thermo-mechanical analgesia method reduce pain intensity in LMWH applications via SC .

SC injection applications are an important part of drug applications and are frequently performed by nurses in clinical practice. Complications resulting from these applications cause physical and mental trauma in patients, they are reluctant to make the next injection, and for nurses, ecchymosis, hematoma and pain occurring at the injection site play a restrictive role in the selection of the site. This is an important problem for patients receiving heparin treatment for a long time; It is seen that different cold application methods such as ice application, cooling spray and thermo-mechanical analgesia techniques are used in heparin injections by SC route. However, there is no study on which these methods are used together and the effects of these methods are compared. This work; The aim of this study was to investigate the effect of three different cold application methods on ecchymosis and pain formation at the injection site in patients undergoing LMWH injection via SC.

ELIGIBILITY:
Inclusion Criteria:

* The patient is 18 years or older,
* Planning LMWH treatment by SC twice a day,
* Has the physical and mental competence to correctly evaluate the Visual Analog Scale (VAS),
* Platelet value is 100 000 / mm³ and ↑
* Prothrombin time (INR) is between 0.87-1.20,
* aPTT value between 22-36 (Platelet, PT and aPTT tests were evaluated considering the reference values of the kits used in the hospital)
* No coagulation disorder,
* Not using oral anticoagulants,
* No scar tissue, incision, lipodystrophy or signs of infection on the skin of the abdomen to be injected,
* No history of cold allergy,
* Agree to participate in the research

Exclusion Criteria:

* Patients who do not agree to participate in the study or who give up during the study and are discharged before the follow-up of SC injection activities will not be included in the sample.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Effects Of Ice Application On Pain In Patients Undergoing Subcutaneous Anticoagulant Therapy | 5 day
  According to the randomization result;
  * Buzzy, a thermomechanical-analgesia device, was placed 30 seconds before the injection in the right upper abdominal region, and the SC injection was applied by sliding the device to the side of the selected region during the injection (Thermomechanical-Analgesia Group),
  * SC-LMWH injection was applied to the right lower abdominal region without any cold application (Control Group),
  * Local coolant spray was applied to the left upper abdominal region from a distance of 15 cm for 5 seconds (Local coolant spray group) and
  * Before and after the application to the left lower abdominal region, the cold application was performed with a cool-pack for 5 minutes (Cool-pack group).
  It was used to evaluate the pain intensity of the patients during and after SC injection. The patient was asked to indicate the pain intensity on a scale immediately after the SC injection and on the 24th, 48th, and 72nd hours after the injection.
Effects Of Ice Application On Ecchymosis In Patients Undergoing Subcutaneous Anticoagulant Therapy | 5 day
  It is a transparent measurement tool designed to measure the size of the ecchymosis formed in the SC injection site, in millimeters. Ecchymosis size was measured with the "Optite-Flexigrid Measurement Tool" in the ecchymoses formed in the 24th, 48th, and 72nd hours after SC-LMWH injection.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Unıversıty- Cerrahpaşa, Şişli, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP, ICF, CSR

REFERENCES:
- [Result] Sendir M, Buyukyilmaz F, Celik Z, Taskopru I. Comparison of 3 methods to prevent pain and bruising after subcutaneous heparin administration. Clin Nurse Spec. 2015 May-Jun;29(3):174-80. doi: 10.1097/NUR.0000000000000129. PMID 25856035
- [Result] Akbari Sari A, Janani L, Mohammady M, Nedjat S. Slow versus fast subcutaneous heparin injections for prevention of bruising and site-pain intensity. Cochrane Database Syst Rev. 2014 Jul 18;(7):CD008077. doi: 10.1002/14651858.CD008077.pub3. PMID 25036897
- [Result] Collado-Mesa F, Net JM, Arheart K, Klevos GA, Yepes MM. Application of a topical vapocoolant spray decreases pain at the site of initial intradermal anaesthetic injection during ultrasound-guided breast needle biopsy. Clin Radiol. 2015 Sep;70(9):938-42. doi: 10.1016/j.crad.2015.04.013. Epub 2015 Jul 7. PMID 26162573
- [Result] Palese A, Aidone E, Dante A, Pea F. Occurrence and extent of bruising according to duration of administration of subcutaneous low-molecular-weight heparin: a quasi-experimental case-crossover study. J Cardiovasc Nurs. 2013 Sep-Oct;28(5):473-82. doi: 10.1097/JCN.0b013e3182578b87. PMID 22760174
- [Result] Mohammady M, Janani L, Akbari Sari A. Slow versus fast subcutaneous heparin injections for prevention of bruising and site pain intensity. Cochrane Database Syst Rev. 2017 Nov 1;11(11):CD008077. doi: 10.1002/14651858.CD008077.pub5. PMID 29090459
- [Result] Cengiz Z, Ozkan M. Comparison of abdominal and arm areas in patients receiving subcutaneous heparin in terms of development of pain, hematoma, and ecchymosis. J Vasc Nurs. 2018 Dec;36(4):208-215. doi: 10.1016/j.jvn.2018.06.003. Epub 2018 Jul 10. PMID 30458944
- [Result] Zaybak A, Khorshid L. A study on the effect of the duration of subcutaneous heparin injection on bruising and pain. J Clin Nurs. 2008 Feb;17(3):378-85. doi: 10.1111/j.1365-2702.2006.01933.x. Epub 2007 Oct 11. PMID 17931375
- [Result] Kuzu N, Ucar H. The effect of cold on the occurrence of bruising, haematoma and pain at the injection site in subcutaneous low molecular weight heparin. Int J Nurs Stud. 2001 Feb;38(1):51-9. doi: 10.1016/s0020-7489(00)00061-4. PMID 11137723
- [Result] Balci Akpinar R, Celebioglu A. Effect of injection duration on bruising associated with subcutaneous heparin: a quasi-experimental within-subject design. Int J Nurs Stud. 2008 Jun;45(6):812-7. doi: 10.1016/j.ijnurstu.2007.02.005. Epub 2007 Mar 30. PMID 17399715
- See also: PREVENTION OF PAIN, BRUISE AND HEMATOMA ON SUBCUTANEOUS HEPARIN INJECTION: A SYSTEMATIC REVIEW — http://www.researchgate.net/publication/319202081_SUBKUTAN_HEPARIN_UYGULAMALARINDA_AGRI_EKIMOZ_VE_HEMATOMUN_ONLENMESI_SISTEMATIK_INCELEME